CLINICAL TRIAL: NCT00421759
Title: Noise-Enhanced Sensory Function in Elders at Risk for Falls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Hyun Gu Kang, PhD, Applied Biodynamics Laboratory, Boston University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG0072; 5P01AG004390-230014; 5P01AG004390 (NIH)
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2008-08

CONDITIONS: Aging; Somatosensory Deficit
Keywords: Sensory loss; psychomotor function; balance; gait

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 85 elderly individuals with somatosensory deficits
  Interventions: Device: Vibrating Insoles
- 2 (Experimental): 85 elderly individuals with recurrent falls
  Interventions: Device: Vibrating Insoles

INTERVENTIONS:
Device: Vibrating Insoles — Participants wear vibrating sandals for 3 trials of 6 minutes, during a single lab visit. The sandal vibration is on during either first or second 3 minutes of the 6 minute trial, as they walk. Also, participants wear the sandals for 2 hours while sitting, with vibrations on for one visit and off for the other.

SUMMARY:
The long-term goal of this project is to develop a non-invasive, noise-based technique for enhancing somatosensation and thereby improving balance control in elderly fallers and older adults with somatosensory deficits.

DETAILED DESCRIPTION:
Previous studies have shown that sub-sensory mechanical noise (i.e., random vibration with a small intensity) can enhance somatosensory function in healthy individuals and older adults with somatosensory deficits. Moreover, the postural sway of both healthy young and healthy elderly individuals during quiet standing can be significantly reduced by applying sub-sensory mechanical noise to the feet using vibrating shoe insoles.

The specific aims of this project are to determine the effects of noise-enhanced somatosensation at the feet on balance performance in elderly individuals with somatosensory deficits and/or recurrent falls, and to assess whether adaptation occurs in noise-enhanced balance control in these individuals. To accomplish these aims, quiet-standing and dynamic posture studies and clinical balance assessments will be conducted on elderly individuals with somatosensory deficits and elderly individuals with recurrent falls (two or more falls over a 12-month period).

This project could lead to the development of a novel bioengineering technique for improving balance control in older adults and patients with somatosensory deficits. The work could thus serve to reduce the frequency, morbidity and cost of falling, and assist aged individuals in achieving maximal independence in activities of daily living and mobility.

Two groups of participants will be recruited from the RNH Epidemiology Core: 85 elderly individuals with somatosensory deficits, and 85 elderly individuals with recurrent falls. The study consists of three visits--a one-hour neurological exam, and two 6-hour laboratory testing sessions scheduled one week apart.

ELIGIBILITY:
Inclusion Criteria:

* Participant must (1) have somatosensory deficit (mild to moderate sensory loss on the bottom of both feet) OR (2) be classified as a recurrent faller (two or more incident falls over a twelve-month period not related to syncope, major medical events, or overwhelming external hazards)
* Age 70 and older
* Able to stand unassisted for at least 60 seconds several times over a 30-minute period
* Able to walk without assistance from a walking aid

Exclusion Criteria:

* Known history of seizures or fainting
* Unstable medical condition
* Open lesions or poor skin condition on feet
* Unable to cooperate with or understand the protocol
* Foot size larger or smaller than the constructed vibrating insoles (men's sizes smaller than 3 or larger than 12; women's sizes smaller than 4.5 or larger than 13.5)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Area ellipse of sway | Three 6-minute trials in one visit, repeated one week later
Berg Functional Balance Scales | Three 6-minute trials in one visit, repeated one week later
Timed Up and Go (TUG)Test | Three 6-minute trials in one visit, repeated one week later
Timed one-legged stance test | Three 6-minute trials in one visit, repeated one week later
Gait timing variability | Three 6-minute trials in one visit, repeated one week later

SECONDARY OUTCOMES:
Changes in: stabilogram-diffusion analysis (SDA) | Three 6-minute trials in one visit, repeated one week later
Neurological risk factors related to falls | Three 6-minute trials in one visit, repeated one week later

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Biodynamics Laboratory, Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Priplata AA, Niemi JB, Harry JD, Lipsitz LA, Collins JJ. Vibrating insoles and balance control in elderly people. Lancet. 2003 Oct 4;362(9390):1123-4. doi: 10.1016/S0140-6736(03)14470-4. PMID 14550702
- [Background] Kiemel T, Oie KS, Jeka JJ. Multisensory fusion and the stochastic structure of postural sway. Biol Cybern. 2002 Oct;87(4):262-77. doi: 10.1007/s00422-002-0333-2. PMID 12386742
- [Background] Laughton CA, Slavin M, Katdare K, Nolan L, Bean JF, Kerrigan DC, Phillips E, Lipsitz LA, Collins JJ. Aging, muscle activity, and balance control: physiologic changes associated with balance impairment. Gait Posture. 2003 Oct;18(2):101-8. doi: 10.1016/s0966-6362(02)00200-x. PMID 14654213
- [Background] Liu W, Lipsitz LA, Montero-Odasso M, Bean J, Kerrigan DC, Collins JJ. Noise-enhanced vibrotactile sensitivity in older adults, patients with stroke, and patients with diabetic neuropathy. Arch Phys Med Rehabil. 2002 Feb;83(2):171-6. doi: 10.1053/apmr.2002.28025. PMID 11833019
- [Background] Priplata A, Niemi J, Salen M, Harry J, Lipsitz LA, Collins JJ. Noise-enhanced human balance control. Phys Rev Lett. 2002 Dec 2;89(23):238101. doi: 10.1103/PhysRevLett.89.238101. Epub 2002 Nov 13. PMID 12485044